Protocol title: Non-invasive Evaluation of Portal
Hypertension in Patients With Compensated
Advanced Chronic Liver Disease by Liver Stiffness
Measurement Using Liver Incytes

PI: Samer Gawrieh, MD

NCT04576897

**Statistical Considerations** 

Document Date: August 5, 2021

Descriptive statistics such as mean, standard error, and percentages were used to characterize the cohort. Comparisons will be made between groups by using Student t test or analysis of variance. Pearson correlation coefficient will be used to detect the correlation between continuous variables. Multivariate analysis will be performed to examine the independent association between dependent and several independent variables. The diagnostic accuracy of LSM will be calculated using area under the receiver operator curve analysis. Sample size is based on clinical experience and precedent established for studies of similar design.